CLINICAL TRIAL: NCT04683887
Title: Randomized and Controlled Prospective Study on Use of the Adhesive Elastic Tape to Control Hand Edema in Patients With a Wrist Fracture Treated With Forearm Plaster.
Brief Title: Taping to Control Edema in Patients With Forearm Plaster for Wrist Fracture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Massimo Guasconi, RN, MSN, Azienda Unita Sanitaria Locale di Piacenza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TapeK_Gesso_ABM_PSO
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Edema Arm; Fracture; Wrist
Keywords: tape; forearm cast
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data processing will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tape application (Experimental)
  Interventions: Device: Tape application
- No tape application (No Intervention)

INTERVENTIONS:
Device: Tape application — Application of the tape with lymphatic technique to the fingers, both dorsally and volarly, of wrist fractured patients treated with a forearm cast
  Arms: Tape application

SUMMARY:
Wrist fractures are a very common event affecting patients of all ages and are estimated to account for approximately 10% -25% of all fractures. 70-90% of fractures are treated with closed reduction and forearm cast. In 2019, 17.4% of wrist fractured patients treated with a plaster cast at the Orthopedic Emergency Department (OED) of the Local Health Unit ("Azienda Unità Sanitaria Locale", AUSL) of Piacenza had a second access to the OED for edema, pain or "intolerance to the plaster cast ".

In literature, there are several studies that demonstrate the effectiveness of adhesive elastic tape for edema control, mostly lymphedema secondary to breast cancer or post-operative edema after knee arthroplasty, although a definitive evidence is still needed.

With this trial, the investigators aim to evaluate the tape effectiveness in counteracting hand edema formation in wrist fractured adult patients treated with forearm cast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with growth plates closed on radiographic examination
* Unilateral distal radius fracture associated or not with ulnar styloid fracture
* Wrist fracture requiring bloodless reduction and immobilization with a forearm cast

Exclusion Criteria:

* Patients with multiple fractures
* Polytrauma patients
* Patients with previous plegia / paralysis of the fractured limb
* Patients with previous lymphedema of the fractured limb
* Patients with access to the OED during the night when the organization does not guarantee the presence of 2 nurses
* Wounds or abrasions in the area of application of the tape
* Acute thrombosis (upper limb veins)
* Scars not perfectly healed in the area of application of the tape
* Dermatitis, psoriatic manifestations or erythema in the area of application of the tape
* Known allergy to acrylic (patch glue)
* Solid neoplasms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic ER o Orthopedic Emergency Department (OED) of the Local Health Unit ("Azienda Unità Sanitaria Locale", AUSL) of Piacenza, Piacenza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guasconi M, Riboni DZ, Granata C, Bolzoni M, Beretta M, Mozzarelli F, Maniscalco P. Randomised controlled prospective study of the use of adhesive elastic tape for the control of hand oedema in patients with a wrist fracture treated in a cast: a study protocol. Int J Orthop Trauma Nurs. 2022 Feb;44:100881. doi: 10.1016/j.ijotn.2021.100881. Epub 2021 Jun 19. PMID 34736885
- [Derived] Guasconi M, Zilli Riboni D, Civardi A, Bolzoni M, Granata C, Beretta M, Genovese A, Mozzarelli F, Quattrini F, Maniscalco P. The use of adhesive elastic tape for hand oedema control in patients with a wrist fracture treated in a cast: A pilot study. Int J Orthop Trauma Nurs. 2024 May;53:101059. doi: 10.1016/j.ijotn.2023.101059. Epub 2023 Oct 22. PMID 38261469

RESULTS

PARTICIPANT FLOW:
Groups:
- No Tape Application: No tape application: Application of the tape will be not done
Period: Overall Study
Arm/Group | Tape Application | No Tape Application
Started | 13 | 10
Completed | 12 | 7
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- No Tape Application: No tape application: Application of the tape not done
- Total: Total of all reporting groups
Arm/Group | Tape Application | No Tape Application | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [67 to 78] | 69 [55 to 72] | 72 [59 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 13 | 10 | 23
Fractured arm [Count of Participants; unit: Participants]
  right | 5 | 3 | 8
  left | 8 | 7 | 15
Number of Participants with Heart diseases [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of Participants with Kidney diseases [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of Participants with Respiratory diseases [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of Participants with Diabetes [Count of Participants; unit: Participants] | 1 | 2 | 3
Number of Participants with Hypertension [Count of Participants; unit: Participants] | 2 | 3 | 5
Thumb circumference at T0 [Median (Inter-Quartile Range); unit: cm] | 7.1 [7.0 to 8.0] | 7.3 [6.7 to 8.0] | 7.1 [6.8 to 8.0]
Circumference of the other 4 fingers (index, middle, ring and pinky) all side by side at T0 [Median (Inter-Quartile Range); unit: cm] | 19.0 [18.0 to 20.2] | 18.0 [16.1 to 18.2] | 18.0 [17.1 to 20.2]
Numerical Rating Scale (NRS) at T0 [Median (Inter-Quartile Range); unit: units on a scale] — Numerical Rating Scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Population: Pain degree at baseline measure was not recorded for 3 subjects of Tape application group and 5 subjects of No tape application group.
  units on a scale
    number analyzed (Participants) | 10 | 5 | 15
    (all) | 5.5 [3.0 to 8.0] | 6.0 [3.0 to 7.0] | 6.0 [3.0 to 8.0]

OUTCOME MEASURES:

1. Primary Outcome: Thumb Circumference
Description: thumb circumference difference between baseline (T0) and follow-up on day 7 (T1)
Time Frame: baseline and 1 week
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Tape Application | No Tape Application
Number analyzed (Participants) | 12 | 7
cm | -0.2 [-0.4 to 0] | 0 [-0.1 to 0.4]

2. Primary Outcome: Circumference of the Other 4 Fingers All Together
Description: difference between T0 and T1 in the circumference of the other 4 fingers (index, middle, ring and pinky) all side by side, measured at the first phalanx
Time Frame: baseline and 1 week
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Tape Application | No Tape Application
Number analyzed (Participants) | 12 | 7
cm | -0.5 [-1.2 to 0] | 0.5 [-0.6 to 0.8]

3. Secondary Outcome: Pain Degree by Numerical Rating Scale (NRS)
Description: pain degree by NRS at T1. The NRS is an 11-point scale used to assess pain intensity, ranging from 0 to 10. A score of 0 indicates no pain, while 10 represents the worst pain imaginable. The NRS is a simple and quick method for patients to self-report their pain level.
Time Frame: 1 week
Population: Pain degree at T1 data is missing for 6 subjects of Tape application group (3 of them also without assessment of NRS at baseline) and 4 subjects of No tape application group (3 of them also without assessment of NRS at baseline).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tape Application | No Tape Application
Number analyzed (Participants) | 6 | 3
score on a scale | 2.5 [1 to 3] | 3 [0 to 4]

4. Secondary Outcome: Number of Participants Taking Painkillers
Description: Number of Participants that have been taken painkillers in the 4 hours prior to T1
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Tape Application | No Tape Application
Number analyzed (Participants) | 12 | 7
Participants | 1 | 0

5. Secondary Outcome: Number of Participants With OED Entry
Description: Number of Participants with at least one OED entry for "intolerance to plaster cast" between T0 and T1
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Tape Application | No Tape Application
Number analyzed (Participants) | 12 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Tape Application | No Tape Application
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7
Other Adverse Events (participants affected / at risk) | 0/12 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT04683887/Prot_SAP_000.pdf